CLINICAL TRIAL: NCT04123340
Title: Intraprocedural Assessment of Ablation Margins Using Computed Tomography Co-registration in Primary Liver Tumor Treatment With Percutaneous Ablation
Acronym: IAMCOMPLETE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Mirada Medical (Unknown)
Responsible Party: Principal Investigator, MCBurgmans, Principal Investigator, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL69217.058.19
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: HCC

STUDY DESIGN:
Intervention Model Description: prospective, single blind, single-arm, phase II stud
Masking Description: post-procedural an assessment will be done of the ablation completeness using registration software. The actual ablation verification will be done qualitatively by the treating physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional intraprocedural CT-scan (Experimental): Additional intraprocedural CT-scan
  Interventions: Diagnostic Test: Additional intraprocedural pre-ablation CT-scan

INTERVENTIONS:
Diagnostic Test: Additional intraprocedural pre-ablation CT-scan — In 20 patients, besides de regular post-RFA scan, a pre-RFA contrast enhanced dual phase CT-scan will be acquired to investigate the feasibility of quantitative ablation assessment.

SUMMARY:
A pre- and postablation scan will be made intraprocedurally to investigate the feasibility of intraprocedural ablation verification assessment using coregistration software

ELIGIBILITY:
Inclusion Criteria:

* Age 18 yrs or above
* HCC very early (0) or early stage (A) according to the BCLC staging system
* Either de novo or recurrent HCC (prior locoregional therapy is allowed in the study)
* Candidate for percutaneous thermal ablation as discussed in a multidisciplinary tumor board. Ablation as 'bridge-to-transplant' is allowed in the study

Exclusion Criteria:

* Estimated GFR <30 ml/min
* Morbid obesitas or any pulmonary condition that is a contraindication to prolonged apnea and high jet-ventilation
* Child Pugh C
* Portal vein tumor invasion
* Extrahepatic metastasis
* Uncorrectable coagulopathy
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Inability or unwillingness to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of the use of co-registration software (>80%) | 1 year
  The proportion of patients in whom reliable co-registration of pre- and post-ablation CT images is feasible

SECONDARY OUTCOMES:
Inter and intra-observer variability | 1 year
  Inter- and intraobserver variability of CT-CT co-registration of determining the minimum ablation margin after thermal ablation for liver tumors
The time that is required for CT-CT co-registration | 1 year
  The time that is required for CT-CT co-registration
Quantitatively assessed ablation margin | 1 year
  Percentage of local recurrence per group as categorized according to ablation margin: <0mm, 0-5mm, >5mm

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
No individual patiend data is shared with researchers.